CLINICAL TRIAL: NCT05677724
Title: Single-cell RNA Sequencing Resolves the Regulatory Role of HBV on the Hepatocellular Carcinoma Immune Microenvironment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fubing Wang (Other)
Responsible Party: Sponsor-Investigator, Fubing Wang, Dr.Prof., Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Other Study IDs: 20220929
Record Dates: First submitted 2022-10-18; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: HBV; Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: HBV DNA(>20000IU/mL)
  Interventions: Diagnostic Test: HBV DNA Sequencing
- Group 2: HBV DNA(>2000IU/mL)
  Interventions: Diagnostic Test: HBV DNA Sequencing
- Group 3: HBV DNA(10-2000IU/mL)
  Interventions: Diagnostic Test: HBV DNA Sequencing
- Group 4: HBV DNA(=<10IU/mL)
  Interventions: Diagnostic Test: HBV DNA Sequencing
- Group 5: HBV DNA(0 IU/mL)
  Interventions: Diagnostic Test: HBV DNA Sequencing

INTERVENTIONS:
Diagnostic Test: HBV DNA Sequencing — Clinical surgical specimens were obtained, cleaned briefly and transported to the laboratory.
  Single-cell suspension preparation and blood cell separation were performed, single-cell sorting suspension was prepared and put on the machine, sorting and library construction were performed, and mRNA sequencing adaptor was docked.
  Single cell data analysis. Based on the findings of single cell analysis, functional verification tests of tumor immune microenvironment cell groups and functional changes of tumor cells were designed.

SUMMARY:
In summary, with the help of single-cell sequencing technology, this study aims to focus on elucidating the influence of HBV-induced hepatocellular carcinoma cell metabolic changes on microenvironment remodeling. With the help of hepatocellular carcinoma microenvironment changes, this study provide a more accurate diagnosis and treatment method for HBV-induced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary liver cancer (hepatocellular carcinoma (HCC)), with evidence of histological or cytological diagnosis, or with HCC meeting conventional clinical diagnostic criteria.
* Both sexes, aged 18-80 years old
* The results of HBVDNA test were in line with the inclusion criteria
* The patient had at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST V1.1)
* Agreed to comply with the study protocol for treatment and follow-up, agreed to provide clinicopathological and follow-up data required by the study, and agreed to use the study data for subsequent research and product development

Exclusion Criteria:

* Other malignant tumors;
* Patients with severe organic diseases do not meet the requirements of infectious liver cancer in this study;
* Suffering from mental illness cannot guarantee the compliance of this study;
* Previous recipients of any cell or organ transplantation;
* Received local regional liver therapy (including various ablations, percutaneous ethanol or acetic acid injections, high-intensity focused ultrasound, transarterial embolization, chemotherapy, or chemoembolization plus embolization) within 14 days prior to study treatment initiation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 patients with primary liver cancer, including 40 single cell sequencing samples (20 cases of liver cancer tissue and 20 cases of paired peripheral blood), were planned to be included and divided into 5 groups. Groups 1-4 were primary liver cancer complicated with hepatitis B infection, and group 5 were hepatitis B negative liver cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical index detection | within 4 hours after the sample was submitted for examination
  HbsAg (IU/mL) \HbsAb (mIU/mL)\HbeAg\HbeAb\HbcAb
HBV DNA copy number | within 24 hours after the sample was submitted for examination
  HBV DNA (IU/mL)
single cell RNA sequencing | within 4 hours after the sample was submitted for examination
  10x genomics chromium 3' sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Fubing Wang, Doctor, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China